CLINICAL TRIAL: NCT07008521
Title: EFFECT OF UNIVERSAL EXERCISE UNIT VERSUS REBOUND THERAPY ON GENU RECURVATUM IN CHILDREN WITH SPASTIC CEREBRAL PALSY
Brief Title: UNIVERSAL EXERCISE UNIT and REBOUND THERAPY ON GENU RECURVATUM Cerebral Palsy Childeren
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Merhan Megahid Hamouda Bakr, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012005355
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-08

CONDITIONS: Genu Recurvatum
Keywords: genu recurvatum, Cerebral Palsy, Universal Exercise Unit, Rebound Therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be assigned randomly into three groups of equal number (control group, study group A and study group B ) the randomization will be performed by simple randomization. Assessors will be blinded to the groups of the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): Control group: Children in this group will receive a traditional physical therapy program.
  Interventions: Procedure: Traditional physical therapy program
- study group A (Experimental): Study group (A): Children in this group will receive a traditional physical therapy program in addition to universal exercise unit program.
  Interventions: Procedure: Universal exercise unit
- Study group B (Experimental): Study group (B): Children in this group will receive the same traditional physical therapy program in addition to rebound therapy
  Interventions: Procedure: Rebound Therapy

INTERVENTIONS:
Procedure: Universal exercise unit — universal exercise unit (UEU) for study groip (A)
  Arms: study group A
Procedure: Rebound Therapy — rebound therpay for study group (B)
  Arms: Study group B
Procedure: Traditional physical therapy program — traditional physical therapy program for contrl group
  Arms: control group

SUMMARY:
to investigate and compare between effectiveness of Universal Exercise Unit and Rebound Therapy on genu recurvatum, muscle strength, balance, functional mobility and quality of life in spastic cerebral palsy children

DETAILED DESCRIPTION:
Children will be equally assigned into three groups using simple randomization, control group, study group (A) and study group (B). Each group will consist of 20 children with spastic CP to overcome any drop out may occur.

Control group: Children in this group will receive a traditional physical therapy program.

Study group (A): Children in this group will receive a traditional physical therapy program in addition to universal exercise unit program.

Study group (B): Children in this group will receive the same traditional physical therapy program in addition to rebound therapy.

Evaluation will be carried out for each child individually before and after 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* -Children with spastic CP both hemiplegic and diplegic.
* Their ages will be ranged from 5-7 years old.
* They will have mild spasticity (grade 1 and 1+) according to Modified Ashworth scale .
* They will be in level I and II according to gross motor function classification system (GMFCS) .
* They will be able to understand orders given to them.

Exclusion Criteria:

* Subjects will be excluded if they have the following:

  1. Visual or hearing impairment.
  2. Severe limb deformities as structural genurecurvatum.
  3. Surgical interference in the lower limbs for the last 6 months.
  4. Botulinum toxin injection of the spastic lower limb muscles during the last six months.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
degree of genu recurvatum | 10 minutes
  degree of genu recurvatum will be measured by Radiological X-Ray

SECONDARY OUTCOMES:
muscle power | 2 minutes
  muscle power will be assessed by using Lafayette Manual Muscle Tester
balance | 20 minutes
  Balance will be assessed by Pediatric Balance Scale
functional mobility | 20 minutes
  Functional mobility will be assessed by Mobility Questionnaire (Mob Quest 28 )
Quality of child life | 20 minutes administration for each child
  Quality of life will be assessed by using Pediatric Quality of Life Inventory (PedsQL) scale

CONTACTS AND LOCATIONS:
Overall Officials: Nanees Essam Mohamed, PhD, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://doi.org/10.1007/s13760-023-02430-8